CLINICAL TRIAL: NCT04500691
Title: pRedicting the Long-term rEsponse of High Frequency sPinal cOrd sTimulation in Patients With Failed Back Surgery Syndrome.
Acronym: REPORT
Status: Completed | Type: Observational
Sponsor: Moens Maarten (Other)
Collaborators: AZ Nikolaas (Other)
Responsible Party: Sponsor-Investigator, Moens Maarten, Principal Investigator, Universitair Ziekenhuis Brussel
Organization: Universitair Ziekenhuis Brussel (Other)
Other Study IDs: REPORT
Record Dates: First submitted 2020-07-09; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Failed Back Surgery Syndrome
Keywords: High frequency Spinal Cord Stimulation; prediction
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FBSS patients: FBSS patients who are treated with high frequency Spinal Cord Stimulation
  Interventions: Other: pain intensity reporting

INTERVENTIONS:
Other: pain intensity reporting — pain intensity reporting

SUMMARY:
The aim of the current retrospective study is to predict responders for HF10-SCS therapy by only using baseline data. Data collected through clinical practice until June 2020 will be used in this retrospective analysis.

ELIGIBILITY:
Inclusion Criteria:

* FBSS patients treated with high frequency spinal cord stimulation implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with FBSS treated with high frequency spinal cord stimulation implantation.
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Responder status | The difference in pain intensity from the date that a patient was eligible for Spinal Cord Stimulation (i.e. baseline) up to the date of the last routine care visit with Spinal Cord Stimulation with database lock at 15th of June 2020.
  A responder is defined as a patient who has 50% pain relief for the predominant pain location at the last follow-up visit compared to baseline.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - UZ Brussel, Jette
  - AZ Nikolaas, Sint-Niklaas